CLINICAL TRIAL: NCT04262752
Title: Automatic Colon-specific Massage With MOWOOT Medical Device to Treat Chronic Constipation in Adults
Brief Title: MOWOOT Device to Treat Constipation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: usMIMA S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOW-01-2017
Record Dates: First submitted 2020-01-31; First posted 2020-02-10 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Constipation; Constipation; Neurogenic; Constipation Chronic Idiopathic
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Each subject in the study will be his/her own control in a BEFORE-AFTER Study, with one group assessed before intervention, during intervention and after intervention.
  Additionally, in order to discuss and analyse the results, further subgroups could be made on the basis of aetiology of the chronic constipation to compare results, i.e.: subjects with constipation derived from Neurogenic Bowel Disease (NBD) vs Idiopathic (No NBD) subjects whose constipation is from unknown origin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronically constipated people (Experimental): Adults with chronic constipation due to either neurogenic bowel dysfunction (NBD) as consequence of a neurogenic condition such as Multiple sclerosis or Parkinson Disease, or to unkwon origin (Idiopathic No-NBD)
  Interventions: Device: intermittent colonic exo-peristaltic massage treatment with the MOWOOT medical device

INTERVENTIONS:
Device: intermittent colonic exo-peristaltic massage treatment with the MOWOOT medical device — The MOWOOT massager belt is connected to the desktop device and is the component which is in contact with the subject giving the abdominal massage action.
  The massager belt, which is placed on the user's abdominal area, administers a specific abdominal massage on the ascendant and descendent segments of the colon. This massage emulates the techniques used by professional therapists through a series of pneumatic actuators operating like the movement of a wave transmitting movement through the colon. The type and speed of the massage can usually be regulated by an algorithm that controls the operation from the desktop device.
  For the present clinical trial, time and force will stay fixed on 20 minutes and force 3 (0'6-0'7 bar). Subjects will not be able to choose other massage options. Subjects should use the MOWOOT device once a day for 20 min (1 complete treatment) ideally at the same hour every day for the 4 weeks of the interventional treatment period.

SUMMARY:
The aim was to assess the safety and effectiveness of the automatic colon-specific massage with the MOWOOT device for patients suffering from chronic constipation due to Multiple Sclerosis, Parkinson Disease (NBD) or other unknown causes (Idiopathic).The hypothesis is that this treatment administered daily in home-use settings could ameliorate constipation in chronically affected people.

DETAILED DESCRIPTION:
The study is an international multi-centre trial using an experimental strategy of once daily abdominal massage using MOWOOT for 4 weeks.

The trial includes a 2-week pre-intervention period with the usual constipation treatment without MOWOOT, followed by a 4-week intervention period consisting of 20 minutes' daily massage with MOWOOT (with or without the usual constipation treatment, as required by subject), followed by 1week wash-out period and finished by 2 weeks' post-intervention follow-up period. The same outcome measures will be assessed before and immediately after the treatment, and again after a washout period.

The principal endpoint of the procedure will be based on constipation improvement (complete bowel movements per week). The secondary endpoints will be based on chronic constipation defined as Rome III criteria assessed by the KESS score, Bristol scale, colonic transit time, dose of laxatives and/or other measures to assist defecation and quality of life. These secondary endpoints regarding defecatory function will be evaluated during intervention and compared with 2 weeks before intervention and 2 weeks after intervention following one week of wash out.

The null hypothesis (H0) is that there is no difference between before and after treatment, against an alternative hypothesis (H1) assuming a difference between the treatments.

Two tailed tests with 95% confidence intervals will be produced for the comparisons of interest in order to investigate the magnitude of treatment effects.

MOWOOT is a "wearable" medical device which emulates the massage techniques used by the professional therapists in order to provide a colon-specific abdominal massage. The product is focused on people who suffer from chronic constipation due to neurogenic bowel disease and prolonged intestinal transit time.

MOWOOT is composed by two main pieces: the desktop device and the massager belt. The desktop device provides the source of energy as well as it contains the panel control which allows the management of the device function and allows to select the treatment time and pressure. The massager belt is connected to the desktop device and is the component which is in contact with the subject giving the abdominal massage action.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil Rome III criteria for functional constipation: include any two of the six symptoms of straining, lumpy or hard stools, sensation of incomplete evacuation, sensation of anorectal obstruction or blockage, digital manoeuvres and less than 3 defecations per week. These should be present during at least 25% of defecations for the last 3 months with symptom onset at least 6 months before the diagnosis;
* Failed routine management of constipation (lack of response to non-stimulant laxatives), or subjects responding to laxative treatment but with secondary diarrhoea and faecal incontinence.
* Duration of constipation more than 6 months.
* If subjects have a diagnosis of multiple sclerosis (MS) or Parkinson disease (PD), it is in a stable phase (no major change in medication for 1 month).
* Subject that have had no abdominal massage for at least 2 months.
* Subjects bothered by their constipation.
* Ability to understand the study
* Ability to come to the outpatient clinic during the study
* Subjects whose constipation aetiology is not only pelvic floor dyssynergia.
* Ability to use MOWOOT or have someone to apply it.
* Subjects that consent to participate in an informed way

Exclusion Criteria:

* Pregnancy or attempt to become pregnant in the next 6 months.
* Subjects alternating constipation and diarrhoea (not due to laxative use)
* Previous large bowel surgery
* The presence of a stoma
* External rectal prolapse
* Active anorexia or bulimia
* Mental inability to give informed consent
* Active abdominal cancer
* Large inguinal or umbilical hernia
* Inflammatory Bowel Disease (IBD)
* Recent abdominal scars, abdominal wounds or skin disorders that may make abdominal massage uncomfortable
* Intra-abdominal implants (catheters, SARS, medication pumps…)
* Subjects already undertaking or have undertaken abdominal massage unless they underwent a previous washout period of at least 2 month.
* Inability to undertake the massage with the device themselves or the lack of a carer willing to do it.
* Participation in another parallel clinical trial or less than 2 month from participation in a previous clinical trial
* Subjects who do not consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Number of complete bowel movements per week | Daily for 9 weeks
  Complete bowel movements mean that the subjects feel they have emptied their bowels completely.

SECONDARY OUTCOMES:
Changes in Constipation symptoms according to the KESS score | Once a week at weeks 2, 6 and 9
  Knowles Eccersley Scott Symptom Score (KESS) is an 11-item questionnaire to diagnose constipation. The assessed items are duration of constipation, laxative use, frequency of bowel movements, unsuccessful evacuatory attempts, feeling incomplete evacuation, abdominal pain, bloating, enemas/digitation, time taken, difficulty evacuation, and stool consistency. Total score ranges from 0 (no symptoms) to 39 (high symptom severity). A cut-off score of ≥ 11 indicates constipation.
Changes in fecal consistency according to Bristol scale | Once a week at weeks 2, 6 and 9
  Bristol stool scale is a worldwide used visual analogue scale that semi-quantitatively assesses faecal consistency from 1 (hard, pellet feces) to 7 (liquid diarrhea). Categories 1 and 2 indicate constipation, 3 and 4 are considered normal, and 5 to 7 indicate soft to liquid feces.
Changes in Colonic transit time (CTT) | Once a week at weeks 2 and 6
  Colonic transit time (CTT) involved the ingestion of 20 radio-opaque markers followed by a single plain abdominal x-ray 5 days later.
Changes in laxative consumption per week | Daily for 9 weeks
  Patients should record on the Bowel diary the names and dose of laxatives, as well as the number of days taking laxatives, among other variables (desire to defecate, number of complete defecations, number of unsuccessful evacuation attempts, painful evacuation, abdominal pain, time taken to evacuate, straining effort, feeling of incomplete evacuation, other symptoms as bloating, influence of constipation on daily activities, need of digital assistance, and concomitant medication)
Changes in other manoeuvres needed to assist defecation per week | Daily for 9 weeks
  Patients should record on the Bowel diary any other manoeuvres needed to assist defecation (such as enemas, digitation, etc.; names and dose) among other variables (desire to defecate, number of complete defecations, number of unsuccessful evacuation attempts, painful evacuation, abdominal pain, time taken to evacuate, straining effort, feeling of incomplete evacuation, other symptoms as bloating, influence of constipation on daily activities, laxatives, and concomitant medication)
Changes in quality of life according to PAC-QoL | Once a week at weeks 2, 6 and 9
  The PAC-QoL is a validated self-reported questionnaire that measures quality of life of subjects with constipation. It is composed of 28 items grouped into four subscales: physical discomfort, psychosocial discomfort, worried and concerns, and satisfaction. Each item is scored from 0 to 4. The lower the score the better quality of life
Changes in subject satisfaction according to a visual analogue scale | Once a week at weeks 2, 6 and 9
  Patients were asked to rate their individual satisfaction with bowel function by answering the question "How do you feel about your defecatory function?" on a visual analogue scale (VAS) from 0 ("No problems to defecate") to 10 ("A lot of problems to defecate").
Adherence to treatment | Once a week during the 4 weeks of the interventional treatment
  The number of completed treatments and the total minutes of each treatment received (completed or not) are automatically registered by the software of the MOWOOT device.

CONTACTS AND LOCATIONS:
Overall Officials: Immaculada Herrero-Fresneda, PhD, Study Chair — usMIMA S.L.; Doreen McClurg, PhD, Principal Investigator — Glasgow Caledonian University
Locations (3):
- Spain (2):
  - Hospital de Terrassa, Terrassa, Barcelona
  - Hospital Universitari MútuaTerrassa, Terrassa, Barcelona
- Glasgow Caledonian University, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Available under demand. Contact with the Chief Scientific Officer of USMIMA S.L by mail: ihf@mowoot.com

REFERENCES:
- [Background] Ayas S, Leblebici B, Sozay S, Bayramoglu M, Niron EA. The effect of abdominal massage on bowel function in patients with spinal cord injury. Am J Phys Med Rehabil. 2006 Dec;85(12):951-5. doi: 10.1097/01.phm.0000247649.00219.c0. PMID 17117000
- [Background] Azpiroz F, Enck P, Whitehead WE. Anorectal functional testing: review of collective experience. Am J Gastroenterol. 2002 Feb;97(2):232-40. doi: 10.1111/j.1572-0241.2002.05450.x. PMID 11866256
- [Background] Bracci F, Badiali D, Pezzotti P, Scivoletto G, Fuoco U, Di Lucente L, Petrelli A, Corazziari E. Chronic constipation in hemiplegic patients. World J Gastroenterol. 2007 Aug 7;13(29):3967-72. doi: 10.3748/wjg.v13.i29.3967. PMID 17663511
- [Background] Coggrave M, Wiesel PH, Norton C. Management of faecal incontinence and constipation in adults with central neurological diseases. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD002115. doi: 10.1002/14651858.CD002115.pub3. PMID 16625555
- [Background] Diego MA, Field T, Hernandez-Reif M, Deeds O, Ascencio A, Begert G. Preterm infant massage elicits consistent increases in vagal activity and gastric motility that are associated with greater weight gain. Acta Paediatr. 2007 Nov;96(11):1588-91. doi: 10.1111/j.1651-2227.2007.00476.x. Epub 2007 Sep 21. PMID 17888059
- [Background] Evans RC, Kamm MA, Hinton JM, Lennard-Jones JE. The normal range and a simple diagram for recording whole gut transit time. Int J Colorectal Dis. 1992 Feb;7(1):15-7. doi: 10.1007/BF01647654. PMID 1588218
- [Background] Harari D, Norton C, Lockwood L, Swift C. Treatment of constipation and fecal incontinence in stroke patients: randomized controlled trial. Stroke. 2004 Nov;35(11):2549-55. doi: 10.1161/01.STR.0000144684.46826.62. Epub 2004 Oct 14. PMID 15486330
- [Background] Knowles CH, Eccersley AJ, Scott SM, Walker SM, Reeves B, Lunniss PJ. Linear discriminant analysis of symptoms in patients with chronic constipation: validation of a new scoring system (KESS). Dis Colon Rectum. 2000 Oct;43(10):1419-26. doi: 10.1007/BF02236639. PMID 11052520
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Liu Z, Sakakibara R, Odaka T, Uchiyama T, Yamamoto T, Ito T, Hattori T. Mechanism of abdominal massage for difficult defecation in a patient with myelopathy (HAM/TSP). J Neurol. 2005 Oct;252(10):1280-2. doi: 10.1007/s00415-005-0825-9. Epub 2005 May 20. No abstract available. PMID 15895308
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] McClurg D, Lowe-Strong A. Does abdominal massage relieve constipation? Nurs Times. 2011 Mar 29-Apr 4;107(12):20-2. PMID 21520798
- [Background] Ng C, Prott G, Rutkowski S, Li Y, Hansen R, Kellow J, Malcolm A. Gastrointestinal symptoms in spinal cord injury: relationships with level of injury and psychologic factors. Dis Colon Rectum. 2005 Aug;48(8):1562-8. doi: 10.1007/s10350-005-0061-5. PMID 15981066
- [Background] Nortvedt MW, Riise T, Frugard J, Mohn J, Bakke A, Skar AB, Nyland H, Glad SB, Myhr KM. Prevalence of bladder, bowel and sexual problems among multiple sclerosis patients two to five years after diagnosis. Mult Scler. 2007 Jan;13(1):106-12. doi: 10.1177/1352458506071210. PMID 17294618
- [Background] Pfeiffer RF. Gastrointestinal Dysfunction in Parkinson's Disease. Curr Treat Options Neurol. 2018 Oct 25;20(12):54. doi: 10.1007/s11940-018-0539-9. PMID 30361783
- [Background] Rao SS, Azpiroz F, Diamant N, Enck P, Tougas G, Wald A. Minimum standards of anorectal manometry. Neurogastroenterol Motil. 2002 Oct;14(5):553-9. doi: 10.1046/j.1365-2982.2002.00352.x. No abstract available. PMID 12358684
- [Background] Ribas Y, Saldana E, Marti-Rague J, Clave P. Prevalence and pathophysiology of functional constipation among women in Catalonia, Spain. Dis Colon Rectum. 2011 Dec;54(12):1560-9. doi: 10.1097/DCR.0b013e31822cb5c2. PMID 22067186
- [Background] Sakakibara R, Yamaguchi C, Uchiyama T, Ito T, Liu Z, Yamamoto T, Awa Y, Yamanishi T, Hattori T. Pelvic autonomic dysfunction without paraplegia: a sequel of spinal cord stroke. Eur Neurol. 2008;60(2):97-100. doi: 10.1159/000138960. Epub 2008 Jun 14. No abstract available. PMID 18552497
- [Background] Sinclair M. The use of abdominal massage to treat chronic constipation. J Bodyw Mov Ther. 2011 Oct;15(4):436-45. doi: 10.1016/j.jbmt.2010.07.007. Epub 2010 Aug 25. PMID 21943617
- [Background] Stewart WF, Liberman JN, Sandler RS, Woods MS, Stemhagen A, Chee E, Lipton RB, Farup CE. Epidemiology of constipation (EPOC) study in the United States: relation of clinical subtypes to sociodemographic features. Am J Gastroenterol. 1999 Dec;94(12):3530-40. doi: 10.1111/j.1572-0241.1999.01642.x. PMID 10606315
- [Background] Su Y, Zhang X, Zeng J, Pei Z, Cheung RT, Zhou QP, Ling L, Yu J, Tan J, Zhang Z. New-onset constipation at acute stage after first stroke: incidence, risk factors, and impact on the stroke outcome. Stroke. 2009 Apr;40(4):1304-9. doi: 10.1161/STROKEAHA.108.534776. Epub 2009 Feb 19. PMID 19228840
- [Background] Talley NJ. Definitions, epidemiology, and impact of chronic constipation. Rev Gastroenterol Disord. 2004;4 Suppl 2:S3-S10. PMID 15184814
- [Background] Ullman T, Reding M. Gastrointestinal dysfunction in stroke. Semin Neurol. 1996 Sep;16(3):269-75. doi: 10.1055/s-2008-1040984. No abstract available. PMID 9085477
- [Background] Winge K, Rasmussen D, Werdelin LM. Constipation in neurological diseases. J Neurol Neurosurg Psychiatry. 2003 Jan;74(1):13-9. doi: 10.1136/jnnp.74.1.13. PMID 12486259
- [Background] Wolters ECh. Non-motor extranigral signs and symptoms in Parkinson's disease. Parkinsonism Relat Disord. 2009 Dec;15 Suppl 3:S6-12. doi: 10.1016/S1353-8020(09)70770-9. PMID 20083010
- [Background] Wood LD, Neumiller JJ, Setter SM, Dobbins EK. Clinical review of treatment options for select nonmotor symptoms of Parkinson's disease. Am J Geriatr Pharmacother. 2010 Aug;8(4):294-315. doi: 10.1016/j.amjopharm.2010.08.002. PMID 20869620
- [Derived] McClurg D, Booth L, Herrero-Fresneda I. Safety and Efficacy of Intermittent Colonic Exoperistalsis Device to Treat Chronic Constipation: A Prospective Multicentric Clinical Trial. Clin Transl Gastroenterol. 2020 Dec;11(12):e00267. doi: 10.14309/ctg.0000000000000267. PMID 33512794